CLINICAL TRIAL: NCT00554853
Title: Peroxisome Proliferator-activated Receptor-gamma Agonists, Rheumatoid Arthritis and Cardiovascular Disease
Brief Title: PPAR-gamma Agonists, Rheumatoid Arthritis and Cardiovascular Disease
Acronym: RAPPAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Mariana Kaplan, Associate Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HUM11806; 5R01HL086553 (NIH)
Record Dates: First submitted 2007-11-06; First posted 2007-11-07 (Estimated); Results first posted 2017-02-02 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2016-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pioglitazone then placebo (Other): Oral daily pioglitazone 30 mg tablets daily for 2 weeks, followed by 45 mg daily tablets until end of study for 3 months compared to placebo in tablets of equal presentation for 3 months, then crossover after a 2 month washout.
  Interventions: Drug: pioglitazone; Drug: Sublingual nitroglycerine
- placebo then study drug (pioglitazone) (Other): Oral daily placebo for 3 months compared to pioglitazone for 3 months, then crossover after a 2 month washout. Similar doses as mentioned above.
  Interventions: Drug: pioglitazone; Drug: Sublingual nitroglycerine

INTERVENTIONS:
Drug: pioglitazone — daily dose, 30 mg daily for 2 weeks followed by 45 mg daily until completing 3 months unless higher dose not tolerated in which case patient remained at 30 mg daily
  Other Names: Actos
Drug: Sublingual nitroglycerine — Used during nitroglycerin-mediated dilatation vascular function measures in both arms of the study if patient's blood pressure permitted. One single tablet was used per vascular test performed.

SUMMARY:
Patients with rheumatoid arthritis have a significantly higher risk to develop heart attacks and other complications of their blood vessels. New therapies are needed to prevent this complication. The purpose of this study is to establish the role of the medication pioglitazone in improving the function of the blood vessels and heart and decreasing the risk of future atherosclerosis development in individuals with rheumatoid arthritis. As a secondary aim-point, we will evaluate the efficacy of pioglitazone in improving rheumatoid arthritis disease activity and markers of inflammation.

DETAILED DESCRIPTION:
This study will establish the role of pioglitazone in improvement of endothelial function, arterial compliance and disease activity in patients with rheumatoid arthritis. This will be a placebo-controlled, double blind, cross-over trial.

Two of the measures which were initially listed as separate outcome measures: (Decrease in inflammation) and Efficacy of pioglitazone in improving rheumatoid arthritis disease activity and markers of inflammation are now shown as a combined score (DAS-28-CRP). The Risks or Side Effects as an outcome measure would be duplicative of the tables in the adverse event section and therefore were deleted as an outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Women on adequate contraception if they are of child-bearing age.
* Meet revised ACR criteria for RA.
* Stable doses of DMARDS,biologic agents and or corticosteroids for at least 3 months.

Exclusion Criteria:

* Pregnant or lactating women.
* Current smokers or individuals who smoked in the last 6 months.
* Diagnosis of Diabetes, heart failure, or infection.
* Current diagnosis of malignant disease except for basal cell or squamous cell carcinoma of the skin.
* No active liver disease.
* No cholesterol-lowering medications or oral hypoglycemic agents.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2007-11; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariana J Kaplan, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Marder W, Khalatbari S, Myles JD, Hench R, Yalavarthi S, Lustig S, Brook R, Kaplan MJ. Interleukin 17 as a novel predictor of vascular function in rheumatoid arthritis. Ann Rheum Dis. 2011 Sep;70(9):1550-5. doi: 10.1136/ard.2010.148031. Epub 2011 Jul 4. PMID 21727237
- [Background] Zhao W, Berthier CC, Lewis EE, McCune WJ, Kretzler M, Kaplan MJ. The peroxisome-proliferator activated receptor-gamma agonist pioglitazone modulates aberrant T cell responses in systemic lupus erythematosus. Clin Immunol. 2013 Oct;149(1):119-32. doi: 10.1016/j.clim.2013.07.002. Epub 2013 Jul 20. PMID 23962407
- [Derived] Marder W, Khalatbari S, Myles JD, Hench R, Lustig S, Yalavarthi S, Parameswaran A, Brook RD, Kaplan MJ. The peroxisome proliferator activated receptor-gamma pioglitazone improves vascular function and decreases disease activity in patients with rheumatoid arthritis. J Am Heart Assoc. 2013 Nov 19;2(6):e000441. doi: 10.1161/JAHA.113.000441. PMID 24252844

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant came into University of Michigan Rheumatology clinic learned about the study and then came in for baseline to sign consent or signed consent at screening visit and then came in for baseline visit at a latter date.
Pre-assignment Details: Out of the 144 individuals screened, one was not randomized to either arm.
Groups:
- Study Drug (Pioglitazone) Then Placebo: Oral daily pioglitazone (study drug for 3 months, followed by 2 month wash out period, then crossover to placebo for 3 months.
- Placebo Then Study Drug (Pioglitazone): Oral daily placebo for 3 months, followed by 2 month wash out period, then crossover to study drug (pioglitazone) for 3 months.
Period: First Arm of Study
Arm/Group | Study Drug (Pioglitazone) Then Placebo | Placebo Then Study Drug (Pioglitazone)
Started | 72 | 71
Completed | 56 | 64
Not Completed | 16 | 7
Period: Washout Period (2 Weeks)
Arm/Group | Study Drug (Pioglitazone) Then Placebo | Placebo Then Study Drug (Pioglitazone)
Started | 56 | 64
Completed | 56 | 57
Not Completed | 0 | 7
Period: Crossover Arm (3 Months)
Arm/Group | Study Drug (Pioglitazone) Then Placebo | Placebo Then Study Drug (Pioglitazone)
Started | 56 | 57
Completed | 53 | 55
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Study Drug (Pioglitazone) Then Placebo: Oral daily pioglitazone for 3 months compared to placebo for 3 months,crossover after a 2 month washout.
- Placebo Then Study Drug (Pioglitazone): Oral daily placebo for 3 months compared to pioglitazone for 3 months, crossover after a 2 month washout.
- Total: Total of all reporting groups
Arm/Group | Study Drug (Pioglitazone) Then Placebo | Placebo Then Study Drug (Pioglitazone) | Total
Number analyzed (Participants) | 72 | 71 | 143
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 59 | 57 | 116
  >=65 years | 13 | 14 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (12.3) | 56.0 (12.0) | 55.2 (12.1)
Gender [Count of Participants; unit: Participants]
  Female | 56 | 53 | 109
  Male | 16 | 18 | 34
Region of Enrollment [Number; unit: participants]
  United States | 72 | 71 | 143

OUTCOME MEASURES:

1. Primary Outcome: Brachial Artery Diameter Change From Baseline in Response to Reactive Hyperemia
Description: This measure represents the percentage change in diameter of brachial artery in response to reactive hyperemia. The data is presented intentionally and only for the results at the conclusion of the study.
Time Frame: 8 months
Population: Vascular function parameters were performed in patients with rheumatoid arthritis at baseline and at completion of each arm , as well as at the beginning of crossover following washout period.
Measure: Mean (Inter-Quartile Range); unit: % changes in diameter of artery
Groups:
- Study Drug (Pioglitazone) Then Placebo: Oral daily study drug (pioglitazone) for 3 months compared to placebo for 3 months, crossover after a 2 month washout.
- Placebo Then Study Drug (Pioglitazone): Oral daily placebo for 3 months compared to study drug (pioglitazone) for 3 months, crossover after a 2 month washout.
Arm/Group | Study Drug (Pioglitazone) Then Placebo | Placebo Then Study Drug (Pioglitazone)
Number analyzed (Participants) | 72 | 71
% changes in diameter of artery | 8.3 [4.4 to 17.5] | 9.43 [4.3 to 20]

2. Secondary Outcome: Rheumatoid Arthritis Disease Activity
Description: Quantification of disease activity using validated assessments (disease activity score on 28 joints (DAS28) and and C-reactive protein ( CRP) (Inflammatory marker) as a combined score (DAS-28CRP)).
  Mean decrease in DAS-28-CRP score when compared to baseline was measured. The range of DAS-28-CRP is 0-10, with 0 meaning no active disease detected and 10 being the most severe active disease detected by joint count and C-reactive protein levels in blood.
Time Frame: 8 mo
Measure: Mean (Standard Deviation); unit: mean decrease in DAS28-CRP score
Groups:
- All Participants While on Placebo: Oral daily study drug (pioglitazone) for 3 months compared to placebo for 3 months, crossover after a 2 month washout.
- All Participants While on Study Drug (Pioglitazone): Oral daily placebo for 3 months compared to study drug (pioglitazone) for 3 months, crossover after a 2 month washout.
Arm/Group | All Participants While on Placebo | All Participants While on Study Drug (Pioglitazone)
Number analyzed (Participants) | 116 | 110
mean decrease in DAS28-CRP score | 0.15 (1.2) | .31 (1.2)
Statistical Analysis 1: Comparison: All Participants While on Placebo vs All Participants While on Study Drug (Pioglitazone); Test type: Superiority or Other; p = 0.63, ANCOVA

ADVERSE EVENTS:
Time Frame: 8 months, but no more than 10 months
Groups:
- Study Drug (Pioglitazone) Then Placebo, While on Drug; Study Drug (Pioglitazone) Then Placebo, During Washout; Study Drug (Pioglitazone) Then Placebo, While on Placebo: Oral daily pioglitazone 45 mg daily(study drug for 3 months, followed by 2 month wash out period, then crossover to placebo for 3 months.
- Placebo Then Study Drug (Pioglitazone) While on Placebo; Placebo Then Study Drug (Pioglitazone) During Washout; Placebo Then Study Drug (Piolglitazone) While on Study Drug: Oral daily placebo for 3 months, followed by 2 month wash out period, then crossover to study drug (pioglitazone) 45 mg daily for 3 months.
Arm/Group | Study Drug (Pioglitazone) Then Placebo, While on Drug | Study Drug (Pioglitazone) Then Placebo, During Washout | Study Drug (Pioglitazone) Then Placebo, While on Placebo | Placebo Then Study Drug (Pioglitazone) While on Placebo | Placebo Then Study Drug (Pioglitazone) During Washout | Placebo Then Study Drug (Piolglitazone) While on Study Drug
Serious Adverse Events (participants affected / at risk) | 5/72 | 1/72 | 0/72 | 1/71 | 3/71 | 5/71
Other Adverse Events (participants affected / at risk) | 22/72 | 2/72 | 8/72 | 12/71 | 0/71 | 9/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Drug (Pioglitazone) Then Placebo, While on Drug (N=72) | Study Drug (Pioglitazone) Then Placebo, During Washout (N=72) | Study Drug (Pioglitazone) Then Placebo, While on Placebo (N=72) | Placebo Then Study Drug (Pioglitazone) While on Placebo (N=71) | Placebo Then Study Drug (Pioglitazone) During Washout (N=71) | Placebo Then Study Drug (Piolglitazone) While on Study Drug (N=71)
Trauma - Car Crash (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Edema, Chest Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspnea, Asthma, Chest Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis - Left Ear (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Right Hip Fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia, Elevated BP (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Infection - Left 1st Toe (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Revision MCP Arthroplasty with Removal of Implant and Rheumatoid Nodule (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
C Diff Colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Breast Cancer (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Intracranial Bleed (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Breast Cancer - Stage 1 (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Low Potassium and Low Sodium Levels (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Death 7 mo post study termination from pneumonia complications of end stage pulmonary fibrosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary Embolus (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Metastic Merkel Cell Cancer (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Drug (Pioglitazone) Then Placebo, While on Drug (N=72) | Study Drug (Pioglitazone) Then Placebo, During Washout (N=72) | Study Drug (Pioglitazone) Then Placebo, While on Placebo (N=72) | Placebo Then Study Drug (Pioglitazone) While on Placebo (N=71) | Placebo Then Study Drug (Pioglitazone) During Washout (N=71) | Placebo Then Study Drug (Piolglitazone) While on Study Drug (N=71)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0 | 0
Weight Gain (Metabolism and nutrition disorders) | 4 | 0 | 0 | 0 | 0 | 0
Swollen, Painful Ankle (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Flushed and Nauseated due to Reaction to Nitroglycerin (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Itchy Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Elevated Blood Pressure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lightheaded (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Decrease Blood Pressure due to Nitroglycerin (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
URI progressed to Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Eczema due to use of Humira (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Left Lower Leg Wound Infection (Cellulitis) (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0
Low Blood Pressure (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0
Headaches (Nervous system disorders) | 3 | 0 | 0 | 3 | 0 | 0
Sprain - Left Knee (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Muscle Aches (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Infection to Salivary Gland (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
RA Flare - Pain in L Wrist and Hand (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Possible Allergic Reaction to Study Drug (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Neck Pain, Cervicalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cervicalgia due to Car Accident (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Infection on the Skin (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Edema / Swelling (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1
Elevated Liver Enzymes (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2 | 0 | 0
Infection of Ulcer on Left 1st Toe (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Edema in the Ankles (Cardiac disorders) | 3 | 0 | 0 | 0 | 0 | 3
Swelling to hands, feet, knees, or legs (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0 | 0 | 0
Bladder Infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 1
Drug Reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hives after Dose Escalation (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Root Canal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 1 | 0 | 0
Tightness in Upper Chest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Shortness of breath (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0
Small Avulsion Right Distal Fibula Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diaphoretic, Low BP (Dehydration), Fainted (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Wheezing (history of Asthma) (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less